CLINICAL TRIAL: NCT06244420
Title: Malignant Myoepithelioma of Bone and Soft Tissues: Diagnostic Imaging and Histology in Relation to Prognosis
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: MYO
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Myoepithelioma
MeSH Terms: conditions — Myoepithelioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: patients with a histological diagnosis of soft tissue or bone malignant myoepithelioma treated from 1998 to 2021.
  Interventions: Other: Clinical data review

INTERVENTIONS:
Other: Clinical data review — review the medical records, radiological imaging, and histological data of these patients

SUMMARY:
The purpose of the study is to assess whether there is a correlation between imaging and histology with prognosis in patients with soft tissue and bone MC from the archives of the Rizzoli Orthopaedic Institute all the patients with a histological diagnosis of soft tissue or bone malignant myoepithelioma treated from 1998 to 2021

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients treated at Rizzoli Orthopaedic Institute between 01 Jan 1998 and 31 Dec 2021
* Age ≥ 2 years old
* Diagnosis of soft tissue or bone malignant myoepithelioma (MC-SB)
* Patients with available clinical and imaging data

Exclusion Criteria:

* At least one inclusion criterion not met

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with soft tissue and bone MC
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation | At baseline (Day 0)
  correlation between imaging and histology with prognosis in patients with soft tissue and bone MC.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Itituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Xu B, Katabi N. Myoepithelial Carcinoma. Surg Pathol Clin. 2021 Mar;14(1):67-73. doi: 10.1016/j.path.2020.09.008. Epub 2021 Jan 5. PMID 33526224
- [Result] Thway K, Fisher C. Myoepithelial tumor of soft tissue: histology and genetics of an evolving entity. Adv Anat Pathol. 2014 Nov;21(6):411-9. doi: 10.1097/PAP.0000000000000039. PMID 25299310